CLINICAL TRIAL: NCT00632073
Title: Effect of Vicriviroc on HIV RNA Levels in Cerebrospinal Fluid
Brief Title: Effect of Vicriviroc on HIV Ribonucleic Acid (RNA) Levels in Cerebrospinal Fluid (Study P05241)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05241
Record Dates: First submitted 2008-01-24; First posted 2008-03-10 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: HIV Infections
Keywords: HIV Infections; Acquired Immunodeficiency Syndrome; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — vicriviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VCV + Failing HAART (Experimental): Vicriviroc plus failing highly-active antiretroviral therapy
  Interventions: Drug: Vicriviroc

INTERVENTIONS:
Drug: Vicriviroc — One tablet of vicriviroc maleate 30 mg once daily for 24 weeks (added to the subject's failing antiretroviral background regimen for 2 weeks, and then administered with optimized background therapy).
  Other Names: Vicriviroc maleate, SCH-D, SCH 417690, VCV

SUMMARY:
Vicriviroc (vye-kri-VYE-rock) is an investigational drug (not yet approved by Government Regulatory Authorities for commercial use) that belongs to a new class of drugs, called CCR5 receptor blockers. This group of drugs blocks one of the ways HIV enters T-cells (the cells that fight infection). Previous studies in HIV treatment-experienced patients have shown that vicriviroc is safe and effective. The purpose of this study is to determine the effect of vicriviroc on HIV RNA levels in cerebrospinal fluid (CSF).

DETAILED DESCRIPTION:
This is a nonrandomized, open-label, multicenter study to investigate the HIV antiviral response in CSF when vicriviroc is added for 2 weeks to the subject's failing antiretroviral background regimen. The primary efficacy endpoint of this study is the mean change in log10 CSF HIV RNA from baseline at Week 2. The secondary efficacy endpoint is the proportion of subjects achieving CSF HIV RNA <50 copies/mL at Week 2. At Week 2, the subject's background regimen will be optimized and vicriviroc continued up to Week 24. After completing Week 24 of the study, subjects will be offered the option to continue on open-label VCV 30 mg once daily, if appropriate, until commercially available or until the sponsor terminates the clinical development of VCV. Subjects who discontinue vicriviroc for any reason will be requested to participate in long-term follow up.

ELIGIBILITY:
Inclusion Criteria:

* A subject must be at least 18 years of age at the time of study entry, of either sex, and of any race.
* A subject must be infected with HIV-1 virus, as documented by a positive assay for HIV-1 RNA in plasma, prior to Screening.
* A subject's HIV isolate must be solely CCR5-tropic at Screening (ie, a subject must not have detectable CXCR4-tropic or dual/mixed CCR5/CXCR4-tropic HIV isolates).
* Subjects must be failing their current antiretroviral regimen with plasma HIV RNA >=1000 copies/mL at the time of screening. (Note: The failing background regimen must contain a ritonavir-boosted PI, and may not include an NNRTI.)
* A subject must be willing to undergo study procedures including lumbar punctures, and to adhere to the chosen antiretroviral regimen.
* A subject must have a pretreatment CSF HIV RNA of >=200 copies/mL.

Exclusion Criteria:

* A subject must not be taking medication for seizure control or have any condition that, in the judgment of the investigator, is likely to increase the risk of seizures.
* A subject must not have a prior history of malignancy (with the exception of surgically resected basal cell carcinoma with clear margins or Kaposi's sarcoma without visceral or mucosal involvement that resolved without systemic anticancer treatment).
* A subject must not have a contraindication to lumbar puncture (eg, bleeding diathesis or use of anticoagulants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change in HIV RNA levels in CSF | Pretreatment and Week 2 visits

SECONDARY OUTCOMES:
Proportion of subjects achieving CSF HIV RNA <50 copies/mL | Week 2